CLINICAL TRIAL: NCT05122286
Title: Randomized Study of Bailout Intracranial Angioplasty Following Thrombectomy for Acute Large Vessel Occlusion: A Multi-centered, Prospective, Open-label, Blind Endpoint, Randomized Controlled Trial (ANGEL-REBOOT)
Brief Title: Randomized Study of Bailout Intracranial Angioplasty Following Thrombectomy for Acute Large Vessel Occlusion
Acronym: ANGEL-REBOOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Zhongrong Miao, Director of Interventional Neuroradiology, Department of Neurology, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HA-X-026(2020)
Record Dates: First submitted 2021-09-25; First posted 2021-11-16 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Acute Ischemic Stroke
Keywords: Endovascular treatment; Large vessel occlusion; Angioplasty; Thrombectomy
MeSH Terms: conditions — Ischemic Stroke | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bailout angioplasty (Experimental): If the patient is randomized into the bailout angioplasty arm, the choice of balloon dilation or stenting will be left to the discretion of the interventionalist.
  Interventions: Procedure: Bailout angioplasty
- Standard therapy (Active Comparator): If the patient is randomized into the standard therapy arm, the interventionalist will decide whether to stop the endovascular recanalization procedure or to perform further recanalization attempts using stent-retrievers and/or aspiration catheters.
  Interventions: Procedure: Standard therapy

INTERVENTIONS:
Procedure: Bailout angioplasty — Use balloons or stents for bailout angioplasty
  Arms: Bailout angioplasty
Procedure: Standard therapy — Stop the endovascular recanalization procedure or to perform further recanalization attempts using stent-retrievers and/or aspiration catheters
  Arms: Standard therapy

SUMMARY:
Unfavorable outcomes were associated with failed thrombectomy of acute large vessel occlusions (LVO). The failed thrombectomy rate was 12-41% reported in multiple randomized controlled trials (RCT). Possible reasons of failed thrombectomy included technical failure of access, failure of retrieving thrombus, thrombotic re-occlusion, and pre-existing intracranial atherosclerotic stenosis (ICAS). Several studies have been published on balloon dilation or permanent stenting as rescue approaches for failed thrombectomy in individual cases, but there is no evidence from RCTs regarding this topic. ANGEL-REBOOT aims to close this gap by performing a randomized study of bailout intracranial angioplasty (balloon dilation and/or stenting) for unsuccessful thrombectomy in LVO patients.

DETAILED DESCRIPTION:
The ANGEL-REBOOT is a multicentered, prospective, randomized, open-label, blinded end-point (PROBE design) study. A total of approximately 348 patients within 24 hours of symptom onset of acute ischemic stroke (NIHSS≥6), who has the imaging evidence of anterior circulation stroke (CT or DWI ASPECTS≥6) or posterior circulation stroke (CT or DWI pc-ASPECTS≥6 and Pons-Midbrain Index [PMI]<3) caused by an occlusion of intracranial internal cerebral artery (ICA), M1 segment of middle cerebral artery (MCA), V4 segment of vertebral artery (VA) or basilar artery (BA).

Randomization would take place after failed thrombectomy (defined as eTICI 0-2a or a remaining high-grade stenosis > 70% after 1-3 attempts of thrombectomy with stent retriever and/or contact aspiration). Patients fulfilling all of the inclusion criteria and none of the exclusion criteria will be randomized 1:1 into two groups (bailout angioplasty or standard therapy) after offering informed content.

If the patient is randomized into the bailout angioplasty arm, the choice of balloon dilation or stenting will be left to the discretion of the interventionalist. If the patient is randomized into the standard therapy arm, the interventionalist will decide whether to stop the endovascular recanalization procedure or to perform further recanalization attempts using stent-retrievers and/or aspiration catheters.

The primary objective is to compare the efficacy and safety of bailout intracranial angioplasty with standard therapy following unsuccessful thrombectomy in acute LVO patients.

The study consists of three visits including 24 hours, 7 days or discharge, and 90 days after randomization. Demographic information, symptoms and signs, laboratory test, neuro-imaging assessment and neurological function scale will be recorded during the study. The primary endpoint is the modified Ranking Scale (mRS) at 90 days. The study is anticipated to last from December 2021 to September 2023 with 348 participants recruited form about 40 centers in China. All the related investigative organization and individuals will obey the Declaration of Helsinki and regulation of Chinese Good Clinical Practice. A scheduled Data and Safety Monitoring Board (DSMB) meeting will oversight the safety and data quality of the study. The trial has been approved by Institutional Review Board (IRB) and Ethics Committee (EC) in Beijing Tiantan hospital, Capital Medical University.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Inclusion criteria

  1. Age ≥18 years
  2. Pre-stroke mRS 0~2
  3. Acute ischemic stroke (NIHSS ≥ 6)
  4. Time-last-known-well to puncture ≤ 24 hours
  5. Informed consent
* Baseline Imaging Inclusion Criteria

  1.Anterior circulation stroke: CT or DWI ASPECTS ≥ 6; Posterior circulation stroke: CT or DWI pc-ASPECTS ≥ 6 and Pons-Midbrain Index (PMI)<3
* Angiographic Inclusion Criteria

  1. Acute ischemic stroke caused by LVO, including intracranial internal cerebral artery (ICA), M1 of the middle cerebral artery (MCA), V4 of vertebral artery (VA) or basilar artery (BA)
  2. Failed recanalization (eTICI 0-2a) or residual severe stenosis (> 70%) after 1-3 attempts of thrombectomy with stent retriever and/or contact aspiration
  3. Microcatheter can pass through the occluded segment before randomization
  4. Occluded artery amenable to angioplasty by judgement of the treating neurointerventionalist

Exclusion Criteria:

1. Any sign of intracranial hemorrhage on brain imaging prior to thrombectomy
2. CT or MRI evidence of mass effect or intracranial tumor
3. Any sign of intracranial vessel perforation during mechanical thrombectomy prior to randomization
4. Contraindication of anti-platelet treatment
5. History of contraindication for contrast medium
6. Current use of oral anticoagulants (e.g. INR > 1.7 for Vitamin K antagonists)
7. Current pregnant or breast-feeding
8. Known to have dementia or psychiatric disease unable to complete neurological assessment and follow-up
9. Life expectancy is less than 3 months
10. Enrolled in another drug or device trial or expected to participate in another drug or device treatment trial within the following 3 months.
11. Any other condition (in the opinion of the site investigator) that inappropriate to participate this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2021-12-19 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Clinical outcome 90 (±14) days after randomization on the modified Ranking Score (mRS) as an ordinal scale (shift analysis) | 90±14 days after randomization
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6 with "0" being perfect health without symptoms to "6" being death.
  Score 0: No symptoms. Score 1: No significant disability. Able to carry out all usual activities, despite some symptoms.
  Score 2: Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  Score 3: Moderate disability. Requires some help, but able to walk unassisted. Score 4: Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  Score 5: Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  Score 6: Dead

SECONDARY OUTCOMES:
Rate of good functional outcome (mRS 0-2) at 90 (±14) days after randomization | 90±14 days after randomization
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6 with "0" being perfect health without symptoms to "6" being death.
  Score 0: No symptoms. Score 1: No significant disability. Able to carry out all usual activities, despite some symptoms.
  Score 2: Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  Score 3: Moderate disability. Requires some help, but able to walk unassisted. Score 4: Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  Score 5: Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  Score 6: Dead
Rate of independent ambulation (mRS 0-3) at 90 (±14) days after randomization | 90±14 days after randomization
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6 with "0" being perfect health without symptoms to "6" being death.
  Score 0: No symptoms. Score 1: No significant disability. Able to carry out all usual activities, despite some symptoms.
  Score 2: Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  Score 3: Moderate disability. Requires some help, but able to walk unassisted. Score 4: Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  Score 5: Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  Score 6: Dead
Functional health status and quality of life (EQ-5D-5L) at 90 (±14) days after randomization | 90±14 days after randomization
  EQ-5D-5L is a standardized instrument for measuring the general health status. Rated level can be coded as a number 1, 2, 3, 4 or 5, which indicates having no problems for 1, having some problems for 2, having moderate problems for 3, having serious problems for 4 and having extreme problems for 5.
Technical success defined as successful recanalization (eTICI 2b-3) of the occluded vessel at the end of the procedure | The end of the procedure
  In brief, eTICI grade 0 is equivalent to no reperfusion or 0% filling of the downstream territory; eTICI 1 reflects thrombus reduction without any reperfusion of distal arteries; eTICI 2a is reperfusion in less than half or 1-49% of the territory; eTICI 2b50 is 50-66% reperfusion, exceeding the modified TICI (mTICI) 2B threshold but below the original TICI 2B cut-off point; eTICI 2b67 is 67-89% reperfusion, exceeding TICI but below TICI 2C; eTICI 2c is equivalent to TICI 2C or 90-99% reperfusion; and eTICI 3 is complete or 100% reperfusion, tantamount to TICI 3.
Infarct volume on FLAIR/T2WI or CT after 18-36 hours of randomization | 18-36 hours after randomization
  The infarct volume is determined on FLAIR or T2-weighted MRI (preferred) or CT if MRI is not feasible.
NIHSS score at 24 hours after randomization | 24 hours after randomization
  The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patent's ability to answer questions and perform activities. Ratings for each item are scored with 3 to 5 grades with 0 as normal, and there is an allowance for untestable items. The single patient assessment requires less than 10 minutes to complete. The evaluation of stroke severity depends upon the ability of the observer to accurately and consistently assess the patient.
Proportion of target vessel recanalization at 18-36 hours after randomization | 18-36 hours after randomization
  Target vessel recanalization defined as grade 2-3 of arterial occlusive lesion (AOL) scale.
  Definition of AOL grades:
  Grade 0--Complete occlusion of the target artery; Grade 1--Incomplete occlusion or partial local recanalization at the target artery with no distal flow; Grade 2--Incomplete occlusion or partial local recanalization at the target artery with any distal flow; Grade 3--Complete recanalization and restoration of the target artery with any distal flow.
Symptomatic intracranial hemorrhage (SICH) defined as the Heidelberg classification within 18-36 hours of randomization | 18-36 hours after randomization
  Heidelberg standard was defined as new intracranial hemorrhage detected by brain imaging associated with any of the item below:
  * 4 points total NIHSS at the time of diagnosis compared to immediately before worsening.
  * 2 point in one NIHSS category. Leading to intubation/hemicraniectomy/ventricular drainage placement or other major medical/surgical intervention.
  * Absence of alternative explanation for deterioration.
Severe procedure-related complications (e.g. dissection of intracranial artery) | 90±14 days after randomization
  Severe procedure-related complications (e.g. dissection of intracranial artery)
Recurrence of ischemic stroke in downstream territory of the occluded vessel within 90 (±14) days after randomization | 90±14 days after randomization
  Recurrence of ischemic stroke in downstream territory of the occluded vessel within 90 (±14) days after randomization
Parenchymal hemorrhage type 2 (PH-2) after 18-36 hours of randomization | 18-36 hours after randomization
  Parenchymal hemorrhage type 2 (PH-2) after 18-36 hours of randomization
Infarct in new territories (INT) within 18-36 hours of randomization | 18-36 hours after randomization
  INT is classified based on two parameters: size (types I, II, and III) and catheter manipulation across territory ostium (types A and B). Thus an INT may be classified as IA, IIB, etc.
  Classification of INT based on size:
  Type I: ≤2 mm diffusion lesion (unidentifiable on CT scan). Type II: >2 mm to ≤20 mm lesion (could potentially be difficult to identify on CT scan).
  Type III: Large (>20 mm) infarct in new territory.
  Classification of INT based on catheter manipulation across territory ostium:
  Type A: Catheter was manipulated past the ostium of the new territory (eg, large ACA infarct in a patient who originally had an M1 occlusion): increased likelihood infarct is related to procedure.
  Type B: Catheter was not manipulated past the ostium of the new territory (eg, left PICA infarct in a patient who originally had a right M1 occlusion): decreased likelihood infarct is related to procedure.
Mortality within 90 (±14) days after randomization | 90±14 days after randomization
  Mortality within 90 (±14) days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Zhongrong Miao, MD, Principal Investigator — Beijing Tiantan Hospital; Feng Gao, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Gao F, Tong X, Wei M, Yao X, Li L, Pan Y, Jia B, Nguyen TN, Yang M, Sun D, Feng G, Yuan G, Xu C, Yuan Z, Wan Y, Wang J, Jing P, Yang X, Wu Z, Hu W, Jiang Y, Wang C, Wen C, Tang J, Luo X, Wu Y, Shen R, Zheng T, Sun Y, Chang M, Liu Y, Haihua Y, Li D, Yin B, Jia W, Wan D, Xu G, Guo Z, Sun D, Wang Y, Duan J, Wang L, Wang G, Wei L, Ma G, Huo X, Mo D, Ma N, Ren Z, Liu L, Zhao X, Wang Y, Fiehler J, Wang Y, Miao Z; ANGEL-REBOOT Study Group. Bailout Intracranial Angioplasty or Stenting After Thrombectomy for Acute Large Vessel Occlusion: 1-Year Outcomes of ANGEL-REBOOT. Circulation. 2025 Nov 18;152(20):1397-1407. doi: 10.1161/CIRCULATIONAHA.125.075429. Epub 2025 Oct 22. PMID 41122847
- [Derived] Li L, Song S, Mo D, Tong X, Miao Z, Gao F; ANGEL-REBOOT Study Group. Factors Associated With Early Reocclusion in Recanalized Intracranial Atherosclerotic Occlusion: ANGEL-REBOOT Insights. Stroke. 2025 Sep;56(9):2431-2439. doi: 10.1161/STROKEAHA.125.051789. Epub 2025 Jun 9. PMID 40485466
- [Derived] Gao F, Tong X, Jia B, Wei M, Pan Y, Yang M, Sun D, Nguyen TN, Ren Z, Demiraj F, Yao X, Xu C, Yuan G, Wan Y, Tang J, Wang J, Jiang Y, Wang C, Luo X, Yang H, Shen R, Wu Z, Yuan Z, Wan D, Hu W, Liu Y, Jing P, Wei L, Zheng T, Wu Y, Yang X, Sun Y, Wen C, Chang M, Yin B, Li D, Duan J, Sun D, Guo Z, Xu G, Wang G, Wang L, Wang Y, Jia W, Ma G, Huo X, Mo D, Ma N, Liu L, Zhao X, Wang Y, Fiehler J, Wang Y, Miao Z. Bailout intracranial angioplasty or stenting following thrombectomy for acute large vessel occlusion in China (ANGEL-REBOOT): a multicentre, open-label, blinded-endpoint, randomised controlled trial. Lancet Neurol. 2024 Aug;23(8):797-806. doi: 10.1016/S1474-4422(24)00186-8. Epub 2024 Jun 21. PMID 38914085
- [Derived] Gao F, Tong X, Jia B, Yang M, Pan Y, Ren Z, Burgin WS, Liu L, Zhao X, Wang Y, Wang Y, Miao Z. Randomised study of bailout intracranial angioplasty following thrombectomy for acute large vessel occlusion (ANGEL-REBOOT): protocol of a multicentre randomised controlled trial. Stroke Vasc Neurol. 2024 Apr 30;9(2):181-188. doi: 10.1136/svn-2023-002433. PMID 37474136